CLINICAL TRIAL: NCT05772741
Title: Grafts of Patient-derived Glioblastoma Stem Cells Onto Autologous Brain Organoids. A Precision Medicine Model for Testing Drugs Against Tumor Invasion
Brief Title: Grafts of GSCs Into Brain Organoids for Testing Anti-invasion Drugs
Acronym: 2253
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Istituto Superiore di Sanità (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2253
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Glioblastoma; Glioma, Malignant
Keywords: glioma stem-like cells; brain organoids; brain invasion; ciliogenesis
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological sample collection (Other): Tumor tissue for glioma stem-like cell culture generation. Skin or PBMC for organoid generation
  Interventions: Other: Biological sample collection

INTERVENTIONS:
Other: Biological sample collection — Collection of biological samples

SUMMARY:
In patients operated for glioblastoma, glioma stem-like cell lines will be obtained from tumor tissue, and IPSCs from skin fibroblasts or PBMCs. Brain organoids will be generated from IPSCs and co-cultured with IPSCs to study brain invasion and ciliogenesis. 3D genome architecture of glioma stem-like cells will be investigated. Gene modulation and pharmacologic strategies to inhibit invasion and restore ciliogenesis will be explored.

ELIGIBILITY:
Inclusion Criteria:

o be enrolled in the study patients must:

1. Have a radiological diagnosis of supratentorial glioblastoma, or
2. Have a radiological diagnosis of first recurrence of a primary supratentorial glioblastoma (for which a formal histopathologic diagnosis of glioblastoma had made at first surgery), according with RANO criteria (Wen, 2010);
3. Be a candidate to neurosurgery for glioblastoma;
4. Be of an age of 18 years or above;
5. Provide written informed consent for participation to the study.

Exclusion criteria

To be enrolled in the study patients must not:

1. Have not enough pathological material removed at surgery available both for mandatory routine histopathological diagnosis and for the present study, as judged by the Principal Investigator;
2. Have not a definitive pathological diagnosis of a primary supratentorial glioblastoma, according with 2016 WHO classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasion | through study completion, an average of 4 years
  Distance travelled by glioma stem cells into brain organoids
Gene assessment | through study completion, an average of 4 years
  Identification of genes responsible of GSC invasion, among those reportedly involved in self-renewal and ciliogenesis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No